CLINICAL TRIAL: NCT02681315
Title: HHHFNC to Prevent Extubation Failure in Preterm Infants: A Randomized Controlled Trial
Brief Title: Comparison of Two Flow Rates of HHHFNC to Prevent Extubation Failure in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University Children Hospital (Other)
Responsible Party: Principal Investigator, Hesham Abdel-Hady, Professor of Pediatrics, Mansoura University Children Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MS/15.10.41
Record Dates: First submitted 2016-02-10; First posted 2016-02-12 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2017-09

CONDITIONS: Prematurity, Mechanical Ventilation
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 6 liter/min group (Experimental): Infants will be extubated to a HHHFNC (Fisher and Paykel Healthcare , Auckland, New Zealand) at ﬂow rate of 6 L/min. Eligible infants will be enrolled while receiving mechanical ventilation. The timing of extubation will be determined by the clinical team and all infants will start caffeine prior to extubation.
  Interventions: Device: HHHFNC 6 liter minute
- 3 liter/min group (Active Comparator): Infants will be extubated to HHHFNC (Fisher and Paykel Healthcare , Auckland, New Zealand) a ﬂow rate of 3 L/min. Eligible infants will be enrolled while receiving mechanical ventilation. The timing of extubation will be determined by the clinical team and all infants will start caffeine prior to extubation.
  Interventions: Device: HHHFNC 3 liters/min

INTERVENTIONS:
Device: HHHFNC 6 liter minute — Infants allocated to HHHFNC at 6 L/min. will be extubated to a HHHFNC flow of 6 L/min. Eligible infants will be enrolled while receiving mechanical ventilation. The timing of extubation will be determined by the clinical team and all infants will start caffeine prior to extubation.
  Arms: 6 liter/min group
Device: HHHFNC 3 liters/min — Infants allocated to HHHFNC at 3 L/min. will be extubated to a HHHFNC flow of 3 L/min. Eligible infants will be enrolled while receiving mechanical ventilation. The timing of extubation will be determined by the clinical team and all infants will start caffeine prior to extubation.
  Arms: 3 liter/min group

SUMMARY:
This is a randomized controlled trial (RCT) to evaluate the influence of two flow rates (6 liter/min versus 3 liter/min) of Heated-Humidified High-Flow-Nasal-Cannula (HHHFNC) on rates of extubation failure in mechanically ventilated preterm infants.

DETAILED DESCRIPTION:
HHHFNC has been proposed as an alternative to nasal continuous positive airway pressure (nCPAP) in neonatal intensive care units (NICUs) for preventing extubation failure. In a recent international survey on periextubation practices in extremely preterm infants, nCPAP was the most common type of respiratory support used (84%) followed by nasal intermittent positive pressure ventilation (55%) and HHHFNC (33%). Moreover, HHHFNC appears to have efficacy and safety similar to those of nCPAP when applied immediately post-extubation to prevent extubation failure in preterm infants. and resulted in significantly less nasal trauma in the first 7 days post-extubation than nCPAP. However, the best flow rates of HHHFNC to prevent extubation failure remains to be known.

This RCT aims to compare the efficacy and safety of postextubation respiratory support via HHHFNC at two different flow rates (6 L/min. versus 3 L/min) regarding successful extubation after a period of endotracheal positive pressure ventilation. We hypothesized that postextubation respiratory support via HHHFNC at a flow rate of 6 L/min. will result in a greater proportion of preterm infants being successfully extubated after a period of endotracheal positive pressure ventilation compared with HHHFNC at a flow rate of 3 L/min.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at less than 37 weeks' gestation, required endotracheal intubation and positive pressure ventilation, and are considered ready for extubation by the clinical team. Infants will be enrolled after written informed parental consent is obtained.

Exclusion Criteria:

* Suspected upper airway obstruction, congenital airway malformations, or major cardiopulmonary malformations

Ages: 1 Hour to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Extubation failure | the 7 days after extubation
  Extubation failure criteria will be defined as follows:
  1. Apnea (respiratory pause >20 seconds), more than 6 episodes requiring physical stimulation in 6 hours or 1 requiring intermittent positive pressure ventilation.
  2. Respiratory acidosis with pH <7.25 and Peripheral arterial oxygen saturation (PaCO2) >65 mmHg.
  ( >15% sustained increase in FiO2 from extubation. 4. Cardiovascular collapse (heart rate <60 beats per minute or shock. 5. Persistent marked/severe retractions. Extubation failure will be deemed to occur if any single criterion was met in any one of the 7 days after extubation. The decision to reintubate an infant and mechanical ventilation variables and subsequent extubation attempts after reintubation will be managed at the discretion of the clinical team.

SECONDARY OUTCOMES:
Mortality | within the 96 hour post-extubation period or at any time after with expected average of 5 weeks
  Death within the 96 hour post-extubation period or at any time after randomization.
Total duration of mechanical ventilation | During NICU admission with expected average of 5 weeks
  Total duration of mechanical ventilation during NICU admission
Total duration of oxygen supplementation | During NICU admission with expected average of 5 weeks
  Total duration of oxygen supplementation during NICU admission
Bronchopulmonary dysplasia (BPD) | at 36 weeks' post-menstrual age.
  BPD defined by oxygen requirement at 36 weeks' post-menstrual age.
Severe BPD | at 36 weeks' post-menstrual age.
  Severe BPD defined as oxygen requirement with fraction of inspired oxygen (FiO2) >0.30 or need for positive pressure support at 36 weeks' post-menstrual age.
The combined outcome variables of death before 36 weeks PMA or BPD | at 36 weeks' post-menstrual age.
  The combined outcome variables of death before 36 weeks PMA or BPD will be used to adjust for occurrence of death after extubation but before the time of assessment of BPD.
The combined outcome variables of death before 36 weeks PMA or severe BPD | at 36 weeks' post-menstrual age
  The combined outcome variables of death before 36 weeks' post-menstrual age (PMA) or severe BPD will be used to adjust for occurrence of death after extubation but before the time of assessment of BPD.
Other neonatal morbidities (intracranial hemorrhage, pneumothorax, patent ductus arteriosus, necrotizing enterocolitis, and retinopathy of prematurity) | baseline, during the 96 hours post-extubation, and at any time thereafter during NICU stay with an expected average of 5 weeks
  The occurrence of neonatal morbidities occurring before, during the 96 hours post-extubation, and at any time thereafter will be documented (intracranial hemorrhage, pneumothorax, patent ductus arteriosus, necrotizing enterocolitis, and retinopathy of prematurity).

CONTACTS AND LOCATIONS:
Overall Officials: Hesham Abdel-Hady, Principal Investigator — Mansoura University Children"s Hospital
Locations (1):
- Neonatal Intensive Care Unit, Mansoura University Children Hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Mandari H, Shalish W, Dempsey E, Keszler M, Davis PG, Sant'Anna G. International survey on periextubation practices in extremely preterm infants. Arch Dis Child Fetal Neonatal Ed. 2015 Sep;100(5):F428-31. doi: 10.1136/archdischild-2015-308549. Epub 2015 Jun 10. PMID 26063193
- [Background] Collaborative Group for the Multicenter Study on Heated Humidified High-flow Nasal Cannula Ventilation. [Efficacy and safety of heated humidified high-flow nasal cannula for prevention of extubation failure in neonates]. Zhonghua Er Ke Za Zhi. 2014 Apr;52(4):271-6. Chinese. PMID 24915914
- [Background] Collins CL, Holberton JR, Barfield C, Davis PG. A randomized controlled trial to compare heated humidified high-flow nasal cannulae with nasal continuous positive airway pressure postextubation in premature infants. J Pediatr. 2013 May;162(5):949-54.e1. doi: 10.1016/j.jpeds.2012.11.016. Epub 2012 Dec 20. PMID 23260098
- [Background] Collins CL, Barfield C, Horne RS, Davis PG. A comparison of nasal trauma in preterm infants extubated to either heated humidified high-flow nasal cannulae or nasal continuous positive airway pressure. Eur J Pediatr. 2014 Feb;173(2):181-6. doi: 10.1007/s00431-013-2139-8. Epub 2013 Aug 18. PMID 23955516